CLINICAL TRIAL: NCT04801602
Title: Comparative Study of Commercially Available Typhoid Point of Care Tests to Benchmark Current and Emerging Tools
Brief Title: Commercial Typhoid Tests Validation Trial
Status: Completed | Type: Observational
Sponsor: Foundation for Innovative New Diagnostics, Switzerland (Other)
Collaborators: Department for International Development, United Kingdom (Other Government)
Responsible Party: Sponsor
Other Study IDs: FE006
Record Dates: First submitted 2021-03-12; First posted 2021-03-17 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Typhoid Fever
Keywords: Typhoid; Enteric Fever; RDTs; Widal test
MeSH Terms: conditions — Typhoid Fever | interventions — Rapid Diagnostic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum samples are stored
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Rapid diagnostic tests — To evaluate different RDTs that are commercially available internationally for detecting antigens or antibodies to Salmonella Typhi and use blood culture as standard for comparison.

SUMMARY:
Typhoid fever (typhoid) is an enteric bacterial infection caused by Salmonella enterica serovar Typhi (Salmonella Typhi; S. Typhi). It is one of the most common bacterial causes of acute febrile illness in the developing world, with an estimated 10.9 million new cases worldwide and 116.8 thousand deaths in 2017. Like many febrile illnesses, typhoid presents with non-specific symptoms and signs, especially in its early stages. In routine healthcare settings in low- and middle-income countries (LMIC), typhoid fever is commonly suspected and treated empirically with antibiotics. This overuse of antibiotics creates a selective pressure for the development of antimicrobial resistance (AMR), that has resulted in the emergence and spread of typhoid strains that are resistant to all first-line antibiotics. Similarly, the low specificity of current rapid diagnostic tests (RDTs) can lead to an over diagnosis of typhoid fever that may result in the overuse of antibiotics and delay the proper treatment for underlying conditions. FIND in collaboration with international typhoid experts developed a target product profile outlining the ideal characteristics of point of care tests. As part of this activity it became apparent that no quality data are available that systematically compare all available commercially point of care tests against the same set of reference standards used in multiple populations (e.g. Africa vs Asia). This lack of benchmarking data significantly impedes health provider's ability to decide on the utility of commercial tests in different settings, ultimately restricting use and access. Further the lack of well characterized samples reduces the ability for targeted innovation in the typhoid space.

The current study aims to benchmark different commercial typhoid tests against a defined reference standard applied in multiple population and simultaneously develop a sample set that can be used in future evaluations of emerging technologies and/or to support innovative test development.

DETAILED DESCRIPTION:
Typhoid is an enteric disease caused by the bacterium Salmonella Typhi; it is estimated that 11 to 20 million people contract typhoid each year and 128 000 to 161 000 die from the disease; children under 5 are at higher risk of contracting the disease.

Typhoid endemic areas are located mainly in South Asia and Sub-Saharan Africa and is transmitted through contaminated water and food. The disease is treatable with a specific antibiotics regimen, however antimicrobial resistance has been reported in several countries, particularly in Pakistan.Several vaccines have been developed but their uptake has been low, partly due to limited information on the exact burden of the disease in endemic countries.

The symptoms of typhoid are similar to other undifferentiated febrile illnesses and typhoid can be mistaken with vector borne febrile illnesses such as scrub typhus.

Blood and bone marrow cultures are considered the gold standard for the diagnosis of typhoid. Those methods require specific infrastructure and skilled staff that are not always available in LMICs and are not adequate for rapid patient management. In addition, although very specific, blood culture sensitivity is impacted by misuse of antibiotics that lower the bacterial load to undetectable levels in patients' blood.

As a consequence, alternatives to blood culture have been used in LMIC. The Widal test is the most used test despite a low performance (sensitivity range: 57-34%; specificity range: 43-83%;reported in several studies. Other options in typhoid diagnosis are rapid diagnostic tests; among them, three tests (Typhidot, Tubex and Test-it™ Typhoid IgM) have been evaluated in several studies. It has been reported a variability of tests performance in different studies and according to the geographical regions. Variability in the test performance reported so far in the literature has hampered WHO to recommend any of these rapid tests in the EDL. FIND in collaboration with international typhoid experts developed a target product profile outlining the ideal characteristics of point of care tests. As part of this activity it became apparent that no quality data are available that systematically compare all available commercially point of care tests against the same set of reference standards used in multiple populations (e.g. Africa vs Asia). These lack of benchmarking data significantly impedes health providers' ability to decide on the utility of commercial tests in different settings, ultimately restricting use and access. Further the lack of well characterized samples reduces the ability for targeted innovation in the typhoid space. A second gap that was identified was the lack of a simple well-performing gold standard suggesting Latent class modelling as a solution used for other pathogens with an imperfect gold standard.

The current study aims to benchmark different commercial typhoid tests against a defined reference standard applied in multiple population and simultaneously develop a sample set that can be used in future evaluations of emerging technologies and/or to support innovative test development.

ELIGIBILITY:
Inclusion Criteria:

* - Individuals aged 8 years of age to 65 years of age
* Body weight equals to or more than 8kgs
* History of fever or axillary temperature of >37.50C for at least 3 consecutive days within the last 7 days prior to enrolment
* Clinical suspicion of enteric fever
* One of the following scenarios:

  * Presents to outpatient department or Emergency Department
  * Admitted to hospital within last 12 hours
* Able and willing to provide informed consent (and assent when required)

Exclusion Criteria:

* Unwillingness to participate in the study

  * Inability to provide the required volume of blood
  * Unwillingness to provide blood
  * Known non-infectious / Non typhoid Infectious causes of fever or other alternate diagnosis of fever
  * Taking anticoagulant drugs
  * Unconscious

Ages: 2 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: The trial population will be composed of adults and children suspected of typhoid between 2-65 years of age. Participants will be recruited when they present to Aga Khan University or its collection site and 3 different hospitals at Nairobi, Kenya
Sampling Method: Probability Sample
Enrollment: 3091 (Actual)
Dates: Start 2020-10-25 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
To evaluate different RDTs that are commercially available internationally for detecting antigens or antibodies to Salmonella Typhi and use blood culture as standard for comparison. | 6-10 months
  Estimates of sensitivity and specificity will be calculated based on the definitions; 95% confidence intervals will be calculated using Wilson's score method.

SECONDARY OUTCOMES:
Establish a biorepository of well characterized specimen collection that can be used to evaluate emerging tests. | 5 years
  does not require any statistical analysis
Evaluation of operational characteristics of different RDTs including invalid and indeterminate rates | 6-10 months
  The number of indeterminate and invalid test results will be reported for each RDT, together with the relative percentage over the total number of tests performed.

CONTACTS AND LOCATIONS:
Overall Officials: Rumina Hasan, M.D, Principal Investigator — AKU; Robert S Onsare, PhD, Principal Investigator — Kenya Medical Research Institute
Locations (2):
- KEMRI, Nairobi, Kenya
- Aga Khan University, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sapkota J, Hasan R, Onsare R, Arafah S, Kariuki S, Shakoor S, Qamar F, Mundalo S, Njeru F, Too R, Ndegwa E, Andrews JR, Dittrich S. Comparative Analysis of Commercially Available Typhoid Point-of-Care Tests: Results of a Prospective and Hybrid Retrospective Multicenter Diagnostic Accuracy Study in Kenya and Pakistan. J Clin Microbiol. 2022 Dec 21;60(12):e0100022. doi: 10.1128/jcm.01000-22. Epub 2022 Nov 30. PMID 36448816